CLINICAL TRIAL: NCT06126601
Title: Incidence and Clinical Impact of Serum Hyperamylasemia (POH) After Pancreatectomy on Postoperative Outcome and Patient Safety
Acronym: HYPPO
Status: Recruiting | Type: Observational
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Sponsor
Other Study IDs: VTG-14; DRKS00031860 (Other: German Clinical Trials Register)
Record Dates: First submitted 2023-08-07; First posted 2023-11-13 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Pancreatectomy; Hyperamylasemia; Pancreatitis, Acute
MeSH Terms: conditions — Hyperamylasemia; Pancreatitis | interventions — Pancreatectomy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Pancreatectomy — Patients who underwent pancreatectomy will be enrolled. Serum amylase and lipase will be measured preoperatively. During surgery, blood samples will be taken after completing the pancreatic anastomosis and at the end of the operation during skin suture. Patients will be followed up during hospital stay, 3 and 6 months after discharge. The clinical outcome (complications, rescue pancreatectomy) will be recorded and analysed.
  Postoperative blood samples, according to clinical standard, will be taken at the 1, 2, 3, 5 and 7 day postoperatively. In addition to amylase several more parameters will be examined intra- and postoperatively: leucocytes, lipase, CRP, bilirubin, transaminases, AP, GGT, creatinine, interleukin-6, PCT. Intraoperative 1-2ml of pancreas juice will be taken for the evaluation of amylase and lipase levels.

SUMMARY:
Recent evidence suggests that postoperative hyperamylasemia (POH) is a predictor of morbidity after pancreatectomy. This is based on the assumption that pancreatitis after pancreatectomy (PPAP) is a major trigger for the development of complications and is indicated by hyperamylasemia. Standardized prospective analysis and correlation with other laboratory parameters, hasn't been performed to date.

Therefore the overall study aims are:

* To prospectively evaluate the incidence and assess the clinical value of biochemical changes for the postoperative course.
* To confirm and improve the definition and classification of postpancreatectomy acute pancreatitis (PPAP) of the International Study Group of Pancreatic Surgery (ISGPS) and to provide knowledge for effective early management of complications.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing pancreatic resection for malignant and benign disease with or without pancreatic anastomosis
* Patients aged 18-85 years
* Willingness to participate as demonstrated by giving a written informed consent.

Exclusion Criteria:

* Necrosectomy (endoscopic or open) for primary acute pancreatitis or within laparotomy
* Age less than 18 years
* Surgical drainage procedures without pancreatic resection (cystojejunostomy for pancreatic pseudocysts)
* One-stage total pancreatectomy
* Missing written consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing a pancreatic resection
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-07-18 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Incidence of PPAP (Postpancreatectomy Acute Pancreatitis) | 90 days after surgery
  Incidence after pancreasresection (pancreatoduodenectomy and distal pancreas resection) according to the definition of ISGPS (International Study Group on Pancreatic Surgery)
Significance of biochemical changes (postoperative hyperamylasemia and hyperlipasemia) | 90 days after surgery
  Correlation with postoperative complications according to the Clavien-Dindo classification and Comprehensive Complication Index ( CCI)

SECONDARY OUTCOMES:
Correlation between hyperamylasemia and rescue pancreatectomy after pancreatoduodenectomy | 90 days after surgery
  Incidence of rescue pancreatectomy after pancreatoduodenectomy with postoperative hyperamylasemia
Correlation between hyperamylasemia and radiological findings for pancreatitis | 90 days after surgery
  Incidence of pancreatitis according to the CT scan postoperatively
Incidence of postoperative mortality | 90 days after surgery
  Postoperative death after complications

CONTACTS AND LOCATIONS:
Overall Officials: Marius Distler, Prof. Dr., Principal Investigator — University Hospital Dresden
Locations (1):
- University Hospital Dresden, Dept. Visceral, Thoracic and Vascular Surgery, Dresden, Germany

IPD SHARING:
Plan to Share IPD: No